CLINICAL TRIAL: NCT07319078
Title: Internet-delivered Psychological Interventions for Pediatric Disorders of Gut-brain Interaction - a Randomised Controlled Study
Brief Title: Pain in Pediatric Patients - Internet Interventions for Disorders of Gut-brain Interaction
Acronym: PIPPI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Ola Olen, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-04544-02
Record Dates: First submitted 2025-12-07; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Irritable Bowel Disease; Functional Abdominal Pain - Not Otherwise Specified (FAP-NOS); Functional Dyspepsia
Keywords: gut-directed hypnotherapy; patient education; disorder of gut-brain intercation; cognitive behavioral therapy; functional abdominal pain; irritable bowel syndrome; randomised controlled trial
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Hypnosis; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: All participants first undergo an online structured patient education program. Thereafter, the participants who still fulfill the diagnostic criteria will be randomised to two treatment arms: 1) internet-delivered cognitive behavioral therapy or 2) gut-directed hypnotherapy via audiofiles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gut-directed hypnotherapy via audiofiles (Experimental): 12-week self-administered hypnotherapy programme. Participants gain access to five different hypnotherapy exercises via audio files and are instructed to listen to them at least once a day.
  Interventions: Behavioral: Gut-directed hypnotherapy
- Internet-delivered cognitive behavioral therapy (Experimental): The participants receive access to a 10-week cognitive behavioral therapy (CBT) -programme.
  Interventions: Behavioral: Cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: Gut-directed hypnotherapy — The programme aims to alleviate gastrointestinal symptoms through deep relaxation and positive suggestions to alter the imagery related to the gut.
  Other Names: Hypnotherapy; Hypnosis; Medical hypnotherapy
  Arms: Gut-directed hypnotherapy via audiofiles
Behavioral: Cognitive-behavioral therapy — The programme is therapist-led and delivered via the internet. It includes exposure-based exercises that aim to improve gastrointestinal symptoms by decreasing avoidance behavior.
  Other Names: CBT; Internet-CBT; Exposure-based CBT
  Arms: Internet-delivered cognitive behavioral therapy

SUMMARY:
Many children and adolescents often experience long-lasting stomach pain. In many cases, this is due to disorders of gut-brain interaction (DGBI), such as irritable bowel syndrome (IBS), functional abdominal pain, and functional dyspepsia. These conditions are caused by disrupted communication between the brain and the gut. They are linked to significant suffering, reduced quality of life, and higher school absenteeism. Psychological treatments such as cognitive behavioral therapy (CBT) have shown good effect, but waiting times within healthcare are often long. Therefore, there is a need for more accessible and cost-effective treatment alternatives.

The goal of this clinical trial is to explore whether gut-directed hypnotherapy, already used successfully in the Netherlands, can be implemented as a new treatment option in Swedish healthcare. In addition, the study will compare gut-directed hypnotherapy with internet-based CBT (iCBT) to learn which digital treatment works best for children and adolescents with DGBI.

Participants will:

Be children or adolescents between 8 and 17 years old.

First take part in a 4-week online education program called the "gut-school," which explains the stomach, the brain, and how symptoms can be managed.

If symptoms remain after the gut-school, be randomly assigned to one of two digital treatments:

iCBT (internet-based cognitive behavioral therapy). 10 week long.

Gut-directed hypnotherapy, delivered as audio recordings to be used at home. 12 week long.

Answer online survey questions before, during, and after treatment so researchers can follow their progress.

These two treatments have never been directly compared. By comparing them, researchers hope to learn not only which treatment works best overall, but also which treatment is most suitable for different participants. The long-term aim is to make gut-directed hypnotherapy, already successful in the Netherlands, available as a treatment option in Sweden.

DETAILED DESCRIPTION:
Gut-directed hypnotherapy has shown promising results in several international studies for the treatment of disorders of gut-brain interaction (DGBI). The treatment builds on relaxation techniques, imagery, and sensory exercises focused on gastrointestinal symptoms. The goal is to improve both awareness of and control over gastrointestinal symptoms. Hypnotherapy is considered safe and has been shown to have very few side effects. International research, particularly from the Netherlands, demonstrates that hypnotherapy leads to better outcomes in both the short and the long term compared to conventional medical treatment. Importantly, home-based audio exercises have been shown to be just as effective as individual face-to-face hypnotherapy delivered by a therapist.

Background and preparation:The research group has already conducted a pilot study in Sweden to test the feasibility of gut-directed hypnotherapy for children with DGBI. In collaboration with Dutch experts, the treatment manual was translated into Swedish, culturally validated by child psychologists, and recorded in high-quality audio format. A secure study platform has been developed to deliver the treatments and collect outcomes, and comprehensive information material for families has been produced, including written texts, films, and audio.

The pilot study, initiated in 2023, showed promising results in the primary outcome measure, PedsQL Gastro, demonstrating improvements in gastrointestinal symptoms. In addition, the pilot provided valuable insights that have led to adjustments in treatment details in order to further optimize the intervention for children and families. These encouraging findings support the implementation of the planned randomized controlled trial and strengthen confidence in the treatment approach, which has now been further optimized based on pilot insights.

Aim: The aim of this randomized controlled trial (RCT) is twofold: first, to evaluate whether gut-directed hypnotherapy can be implemented as a digital treatment option within Swedish healthcare, and second, to compare its effectiveness with internet-based cognitive behavioral therapy (iCBT). These two evidence-based psychological treatments have never before been directly compared. The trial seeks to determine not only which treatment is most effective overall, but also which treatment may be best suited for different participants.

Study population:The RCT will recruit approximately 300 children and adolescents aged 8-17 years who meet diagnostic criteria for DGBI according to the Rome IV classification. Recruitment will take place at pediatric gastroenterology clinics and general pediatric units across Sweden, including both specialized gastroenterology centers and local child health clinics. Before enrollment, all families will talk with a study physician or study nurse to review inclusion and exclusion criteria, receive study information, and go through the principles of both treatment options.

Exposure: All participants will begin with a four-week digital education program called the "gut-school," designed to provide knowledge about the gut-brain interaction and strategies to manage symptoms. Participants who still report symptoms after completing the gut-school, and who are motivated to continue, will be eligible to enter the next phase of the study. These participants will be randomized in a 1:1 ratio to one of two active treatment arms. The hypnotherapy arm will consist of audio-based self-exercises performed at home every day for 12 weeks. The iCBT arm will consist of a structured, therapist-guided internet-based CBT program for abdominal pain, lasting 10 weeks. Both treatments will be delivered through the secure study platform, with the option to access materials via mobile devices.

Outcome: The primary outcome will be change in PedsQL Gastro, a validated questionnaire that measures gastrointestinal symptoms and their impact on daily life and quality of life. A clinically significant improvement will be defined in line with international recommendations. Secondary outcomes will include school attendance, psychological well-being, and health-related quality of life.

All outcomes will be collected both from children and from their parents, using parallel versions of the validated questionnaires. Data will be collected at baseline, every third week during treatment, immediately after completion, and at 6- and 24 months follow up, all through the secure digital platform with identification control.

A comprehensive health economic evaluation will be conducted, adopting a societal perspective to capture all relevant costs and consequences. Resource use will be assessed using the Trimbos and Institute of Technology Cost Questionnaire for Psychiatry (TIC-P), which measures direct medical, non-medical, and productivity-related costs over the preceding four weeks. Health-related quality of life will be assessed using PedsQL, which will be mapped to CHU9D to derive utilities and calculate QALYs (quality-adjusted life years). Both costs and QALYs will be discounted according to standard economic evaluation guidelines. Incremental cost-effectiveness ratios (ICERs) will be computed to compare interventions, and uncertainty will be explored. The analysis will adhere to international standards for trial-based economic evaluations.

Power:The research group has conducted a formal power analysis for the planned RCT. The analysis was based on results from the Swedish pilot study studies in both gut-directed hypnotherapy and cognitive behavioral therapy, including internet-based CBT. With these data as reference, the trial is designed to recruit 300 participants to ensure adequate power to detect clinically meaningful differences between treatment arms. The study is scheduled to run for two years, starting in autumn 2025.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-17 years
* Basic somatic work-up completed (CRP/ESR, TGA, complete blood count, fecal calprotectin)
* Confirmed DGBI diagnosis: IBS, functional abdominal pain, or functional dyspepsia (according to Rome IV criteria)
* Any constipation must be treated according to current clinical guidelines, with stable laxative dosing for at least one month prior to referral
* In cases of celiac disease, the participant must have followed a gluten-free diet for at least six months and TGA values must have normalized
* For participants with a neuropsychiatric diagnosis treated with medication, at least two months must have passed since the last dose adjustment
* At least one parent and the child/adolescent must be fluent in Swedish and willing to participate in both the educational program and treatment (regardless of randomization outcome), complete homework assignments, and respond to questionnaires

Exclusion Criteria:

* Other organic disease that better explains the gastrointestinal symptoms
* At referral assessment, psychiatric symptoms or psychosocial problems - such as severe bullying, high school absenteeism, or difficult family circumstances - are judged to be more prominent than the gastrointestinal problems and require more extensive, multiprofessional care than what the study can offer
* Participants who have already completed gut-directed hypnotherapy or CBT

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Peds QL gastro | Assessments will be collected at baseline, after the gut-school (and before randomization), every third week during treatment (week 3, 6, 9 and 12), and at 6-month follow-up
  Description: Short questionnaire gastrointestinal symptom scale. Minimum value 0, maximum value 100, higher score means better outcome.

SECONDARY OUTCOMES:
Pain frequency | Assessments will be collected at baseline, after the gut-school (and before randomization), every third week during treatment (week 3, 6, 9 and 12), and at 6- and 24- month follow-up.
  Assessed by asking participants how many minutes or hours they have experienced abdominal pain during each day of the same 7-day period. This will give an estimate of the overall duration of pain episodes in addition to their intensity.
Pain intensity | Assessments will be collected at baseline, after the gut-school (and before randomization), every third week during treatment (week 3, 6, 9 and 12), and at 6- and 24- month follow-up.
  Assessed with the Wong-Baker FACES Pain Rating Scale, a validated tool for children. At each measurement point, participants will rate their pain once daily for seven consecutive days, providing a weekly average of pain intensity.
Stress | Assessments will be collected after the gut-school (and before randomization), every third week during treatment (week 3, 6, 9 and 12), and at 6-month follow-up
  PAS pediatric stress questionnare. Minimum value 0, maximum value 44, higher score means worse outcome
Gastrointestinal symtom -related anxiety | Assessments will be collected at baseline, after the gut-school (and before randomization), every third week during treatment (week 3, 6, 9 and 12), and at 6-month follow-up.
  BRQ-C questionnare. Minimum value 11, maximum value 77, higher score means worse outcome.
GI symptom specific anxiety | Assessments will be collected after the gut-school (and before randomization), every third week during treatment (week 3, 6, 9 and 12), and at 6-month follow-up
  VSI: Visceral sensitivity index short scale. Minimum value 0, maximum value 35, higher score means worse outcome.
Quality of life | Assessments will be collected at baseline, after the gut-school (and before randomization), every third week during treatment (week 3, 6, 9 and 12), and at 6-month follow-up
  Peds-QL- QOL. Minimum value 0, maximum value 100, higher score means better outcome.
Adequate relief | Assessments will be collected after the gut-school (before randomization), every third week during treatment (week 3, 6, 9 and 12), and at 6-month follow-up
  SAQ. Minimum value 0, maximum value 7, higher score means better outcome
Self efficacy | Assessments will be collected after the gut-school (and before randomization), every third week during treatment (week 3, 6, 9 and 12), and at 6-month follow-up
  This questionnaire measures how confident a person feels in managing gastrointestinal symptoms, such as abdominal pain, discomfort, or nausea. Confidence is rated on a scale from 0 ("not at all confident") to 100 ("completely confident"). The aim is to capture self-efficacy in handling symptoms without relying on medication.

OTHER OUTCOMES:
Utilisation of health-care resources | The TIC-P will be administered at baseline, post-intervention, and at 6- and 24-month follow-up for both treatment arms (hypnotherapy and internet-based CBT).
  Resource use will be assessed using the Trimbos and Institute of Technology Cost Questionnaire for Psychiatry (TIC-P), which measures direct medical, non-medical, and productivity-related costs over the preceding four weeks. A comprehensive health economic evaluation will be conducted, adopting a societal perspective to capture all relevant costs and consequences.

CONTACTS AND LOCATIONS:
Overall Officials: Ola Olén, Professor, Study Chair — Karolinska Institutet
Locations (1):
- Sachs Children's Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://ki.se/pippi-projektet